CLINICAL TRIAL: NCT06320808
Title: Evaluating FDA's Proposed Patient Medication Information Handout: A Randomized Trial Measuring Perceived Usefulness and Comprehension
Brief Title: Evaluating FDA's Proposed Patient Medication Information Handout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Baruch Fischhoff, University Professor, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY2023_00000449
Record Dates: First submitted 2024-03-08; First posted 2024-03-20 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2024-06

CONDITIONS: Knowledge; Attitude
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either the one-page FDA-template PMI (FDA PMI), a modified template, which added information about drug benefits (Decision Critical PMI), or the existing drug information insert (standard drug information). Participants will complete the same survey questions measuring perceived usefulness and comprehension of the information.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FDA-template PMI (Experimental): Patient medication information designed according to FDA template
  Interventions: Other: FDA template PMI
- Decision Critical PMI (Experimental): Patient medication information designed according to FDA template and modified, according to decision science principles, to include benefit information
  Interventions: Other: Decision Critical PMI
- Standard Information (Experimental): Standard of care patient medication information
  Interventions: Other: Standard Information

INTERVENTIONS:
Other: FDA template PMI — Intervention is an information format viewed by participants. The patient medication information format was designed according to a proposed FDA template, which provides information about safe and effective use of a medication. No drug or device is included as part of this intervention.
  Arms: FDA-template PMI
Other: Decision Critical PMI — Intervention is an information format viewed by participants. The patient medication information format was designed according to a proposed FDA template and modified, according to decision science principles, to include benefit information, which provides information about safe and effective use of a medication. No drug or device is included as part of this intervention.
  Arms: Decision Critical PMI
Other: Standard Information — The intervention is an information format viewed by participants. This patient medication information format is the current standard of care patient medication information that is included with the drug. No drug or device is included as part of this intervention.
  Arms: Standard Information

SUMMARY:
The goal of this study is to assess how useful the proposed one-page FDA-template PMI is to potential users.

The main questions it aims to answer are:

How does the proposed one-page FDA-template PMI compare with the current drug information insert in terms of usefulness and comprehension?

and

How does the proposed one-page FDA-template PMI compare with a revision adding drug benefit information?

Participants will randomized to review one of three patient medication information sheets and then asked questions related to usefulness and comprehension.

DETAILED DESCRIPTION:
The US Food and Drug Administration (FDA) has proposed a new one-page 'patient medication information (PMI) handout that can be provided with every prescription medication, in order to provide patients with the information they need to use their medications safely and effectively. The current proposal omits some decision-critical benefit information and had not been tested with potential users, potentially undermining its effectiveness.

The goal of this study is to assess how useful the proposed one-page FDA-template PMI is to potential users, compared with a revision adding drug benefit information and with the current drug information insert.

A randomized trial will be conducted with U.S. female adults 18-45 years, recruited in March, 2024. Participants will complete an online survey after being randomized to view 1 of the 3 information formats. Participants will be paid $10. Surveys are expected to take no more than 30 minutes to complete.

Participants will be randomized to receive either the one-page FDA-template PMI (FDA PMI), a modified template, which added information about drug benefits (Decision Critical PMI), or the existing drug information insert (standard drug information) for the drug, Mifeprex. All individuals will complete knowledge and usability questions and provide demographic information.

The main outcomes measured will be perceived usefulness and comprehension of the patient medication information.

ELIGIBILITY:
Inclusion Criteria:

* US geographic location
* 18-45 years of age
* assigned female sex at birth

Exclusion Criteria:

* <18 years of age
* > 45 years of age
* assigned a sex other than female at birth

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Limited to females of reproductive age
Enrollment: 330 (Actual)
Dates: Start 2024-03-03 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Perceived difficulty or ease in reading information | day 1
  Single question with a 5-point likert scale response for "How easy or difficult was it to read the medication information guide about [drug]?" Minimum score is 1; Maximum score is 5. A higher score represents higher perceived usefulness.
Perceived usefulness of the medication information guide in making a use decision | day 1
  Single question with a 5-point likert scale response for "For someone who had not yet decided to use [drug], how useful would the medication information guide be in helping them to make that decision?" Minimum score is 1. Maximum score is 5. A higher score represents higher perceived usefulness.
Perceived usefulness of the medication information guide in taking the medication properly | day 1
  Single question with a 5-point likert scale response for "If someone had decided to use [drug], how useful would the medication information guide about [drug] be in helping them use the drug properly? " Minimum score is 1. Maximum score is 5. A higher score represents higher perceived usefulness.
Comprehension | day 1
  10 newly-constructed questions designed to measure the comprehension of the following information from the medication information guide: 1) Analysis of condition (1 question) 2) Risks (3 questions) 3)Risk Management (3 questions), and 5) Benefits (3 questions). Participants can score from 0-10 with 10 representing full comprehension of the information and 0 representing no comprehension of the information.

SECONDARY OUTCOMES:
Strength of Evidence | day 1
  3 questions measuring strength of evidence. One asking about perceived strength of evidence, one about safety, and one about effectiveness of the medication. Each measured on a 5-point likert scale. The question text for each question, respectively, is "how strong is the scientific evidence that [drug], when taken correctly, helps patients [purpose of drug]?" "how safe is [drug], when taken correctly, for [purpose of drug]? "how effective is [drug], when taken correctly, for [purpose of drug]?"

CONTACTS AND LOCATIONS:
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No